CLINICAL TRIAL: NCT05834907
Title: Prevention of Attachment Insecurity, Physiological Dysregulation, and Child Behavior Problems
Brief Title: Hands and Hearts Together
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Lehigh University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jude Cassidy, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1857396-18; 1R01HD105676-01A1 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Parent-Child Relations; Development, Infant; Parenting; Development, Child
Keywords: Parent-Child Relations; Development, Infant; Parenting; Development, Child; Attachment; Home Visiting; Early Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circle of Security Parenting (COS-P) (Experimental): These participants will receive the Circle of Security Parenting (COS-P) intervention, an attachment-based, manualized, 8-session (90 minutes/session), home visiting intervention.
  Interventions: Behavioral: Circle of Security Parenting
- Little Talks (Active Comparator): These participants will receive the Little Talks intervention, a manualized, 8-session (90 minutes/session) early literacy home visiting intervention.
  Interventions: Behavioral: Little Talks

INTERVENTIONS:
Behavioral: Circle of Security Parenting — COS-P is an attachment-based, home visiting intervention intended to supporting parents in serving as "a secure base" from which their children can explore the world, and to which their children can return in times of distress (Bowlby, 1988). Such secure base parenting increases the likelihood of children's secure attachment. COS-P also targets parental responses to children's expression of their needs (e.g., crying), and is designed to help parents understand the ways in which their own (parental) dysregulated emotional, physiological, and behavioral responses to children's emotions and behaviors can limit their responsiveness to their children's attachment needs.
  Arms: Circle of Security Parenting (COS-P)
Behavioral: Little Talks — Little Talks is an early literacy home visiting intervention developed for low-income, racial and ethnic minority infants and toddlers, and has been tested in Early Head Start contexts (Manz et al., 2016; Manz et al. 2017). Little Talks uses book sharing to promote early literacy and has been adapted in both English and Spanish. The intervention utilizes modular treatments during home visits, teaching parents how to facilitate language interactions with their children through book sharing. Age appropriate books are given to parents to share with their children during the intervention.
  Arms: Little Talks

SUMMARY:
Growing evidence demonstrates that secure attachment in childhood predicts children's healthy social, biological, and behavioral functioning, whereas insecure attachment predicts behavior problems and physiological dysregulation; thus, efforts to foster secure attachment are crucial for promoting the healthy development of children and families. This proposal describes a randomized controlled trial (RCT) of an innovative intervention program that can be widely implemented designed to foster children's secure attachment, promote healthy physiological regulation, and reduce the risk for behavior problems: The Circle of Security ® Parenting (COS-P) intervention. To this end, investigators will conduct an RCT with 249 parent-child dyads enrolled or are eligible but not yet enrolled in two diverse Early Head Start (EHS) programs.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children (age 8 to 36 months) are enrolled or are eligible to be enrolled in Harrisburg PA and Lehigh Valley PA Early Head Start programs

Exclusion Criteria:

* Parents who are not sufficiently fluent in the language in which COS-P intervention will be conducted (Spanish or English)

Min Age: 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Strange Situation Procedure (SSP) #1 | Baseline
  Child-parent attachment for children aged 12-24 months will be assessed with Ainsworth's Strange Situation (Ainsworth et al., 1978) procedure. The 20-minute procedure consists of two infant-parent separations, and two reunions. Infant behavior is used to classify infants as secure or one of three types of insecure; continuous security scores can also be derived, and will be used in addition to classifications.
Strange Situation Procedure (SSP) #2 | Immediately post-intervention
  Child-parent attachment for children aged 12-24 months will be assessed with Ainsworth's Strange Situation (Ainsworth et al., 1978) procedure. The 20-minute procedure consists of two infant-parent separations, and two reunions. Infant behavior is used to classify infants as secure or one of three types of insecure; continuous security scores can also be derived, and will be used in addition to classifications.
Strange Situation Procedure (SSP) #3 | 6-month follow up
  Child-parent attachment for children aged 12-24 months will be assessed with Ainsworth's Strange Situation (Ainsworth et al., 1978) procedure. The 20-minute procedure consists of two infant-parent separations, and two reunions. Infant behavior is used to classify infants as secure or one of three types of insecure; continuous security scores can also be derived, and will be used in addition to classifications.
Macarthur Preschool Strange Situation (PACS) #1 | Baseline
  Child-parent attachment for children over 24-months will be assessed with the MacArthur Preschool Strange Situation (PACS; Cassidy et al., 1992; Solomon & George, 2016), which also classifies children as secure or one of three types of insecure; continuous security scores on a scale of 1 to 7 can also be derived, and these (standardized) scores will be used along with classifications. This procedure consists of an initial 3-minute period in which both parent and child are in the toy-filled playroom, followed by two separations (3 and 5 minute) and two 3-minute reunions.
Macarthur Preschool Strange Situation (PACS) #2 | Immediately post-intervention
  Child-parent attachment for children over 24-months will be assessed with the MacArthur Preschool Strange Situation (PACS; Cassidy et al., 1992; Solomon & George, 2016), which also classifies children as secure or one of three types of insecure; continuous security scores on a scale of 1 to 7 can also be derived, and these (standardized) scores will be used along with classifications. This procedure consists of an initial 3-minute period in which both parent and child are in the toy-filled playroom, followed by two separations (3 and 5 minute) and two 3-minute reunions.
Macarthur Preschool Strange Situation (PACS) #3 | 6-month follow up
  Child-parent attachment for children over 24-months will be assessed with the MacArthur Preschool Strange Situation (PACS; Cassidy et al., 1992; Solomon & George, 2016), which also classifies children as secure or one of three types of insecure; continuous security scores on a scale of 1 to 7 can also be derived, and these (standardized) scores will be used along with classifications. This procedure consists of an initial 3-minute period in which both parent and child are in the toy-filled playroom, followed by two separations (3 and 5 minute) and two 3-minute reunions.
Cortisol Stress Reactivity and Recovery #1 | Baseline
  Cortisol stress reactivity and recovery will be assessed (following previous studies; e.g., Luijk et al., 2010) using the Strange Situation Procedure (SSP) as the stressor. Salivary samples will be collected (using a 125mm polymer swab) at baseline (pre-task), 10-, 20-, 30-, and 40-minutes post peak SSP stressor (i.e., end of separation 2), then frozen in tubes. Radioimmunoassay analysis will be done in duplicate, with the mean used as the final measure (in ug/dl). Labs will begin in the afternoon (between 1-4pm) to reduce potential diurnal effects. Multiple studies (e.g., Bernard & Dozier, 2010; Thompson et al., 2015) demonstrated a lack of diurnal influence in infant cortisol studies, thus time of day will not be controlled. Cortisol may fluctuate with sleep/wake patterns and eating (Gunnar & Herrera, 2013), so investigators will control for time of last waking and eating.
Cortisol Stress Reactivity and Recovery #2 | Immediately post-intervention
  Cortisol stress reactivity and recovery will be assessed (following previous studies; e.g., Luijk et al., 2010) using the Strange Situation Procedure (SSP) as the stressor. Salivary samples will be collected (using a 125mm polymer swab) at baseline (pre-task), 10-, 20-, 30-, and 40-minutes post peak SSP stressor (i.e., end of separation 2), then frozen in tubes. Radioimmunoassay analysis will be done in duplicate, with the mean used as the final measure (in ug/dl). Labs will begin in the afternoon (between 1-4pm) to reduce potential diurnal effects. Multiple studies (e.g., Bernard & Dozier, 2010; Thompson et al., 2015) demonstrated a lack of diurnal influence in infant cortisol studies, thus time of day will not be controlled. Cortisol may fluctuate with sleep/wake patterns and eating (Gunnar & Herrera, 2013), so investigators will control for time of last waking and eating.
Cortisol Stress Reactivity and Recovery #3 | 6-month follow up
  Cortisol stress reactivity and recovery will be assessed (following previous studies; e.g., Luijk et al., 2010) using the Strange Situation Procedure (SSP) as the stressor. Salivary samples will be collected (using a 125mm polymer swab) at baseline (pre-task), 10-, 20-, 30-, and 40-minutes post peak SSP stressor (i.e., end of separation 2), then frozen in tubes. Radioimmunoassay analysis will be done in duplicate, with the mean used as the final measure (in ug/dl). Labs will begin in the afternoon (between 1-4pm) to reduce potential diurnal effects. Multiple studies (e.g., Bernard & Dozier, 2010; Thompson et al., 2015) demonstrated a lack of diurnal influence in infant cortisol studies, thus time of day will not be controlled. Cortisol may fluctuate with sleep/wake patterns and eating (Gunnar & Herrera, 2013), so investigators will control for time of last waking and eating.
Child Behavior Checklist (CBCL) #1 | Baseline
  Child behavior problems will are assessed with the Child Behavior Checklist (version for 1.5- to 5-year-olds; CBCL; Achenbach & Rescorla, 2000). Parents will complete this widely used 100-item questionnaire to report their children's internalizing (36 items, e.g., "is nervous, withdrawn") and externalizing (24 items, e.g., "is restless, disobedient") behavior problems. Responses are given on a 3-point scale: (0) not true, (1). somewhat/ sometimes true, (2) very/often true). Items are summed to create subscales for internalizing and externalizing problems.
Child Behavior Checklist (CBCL) #2 | Immediately post-intervention
  Child behavior problems will are assessed with the Child Behavior Checklist (version for 1.5- to 5-year-olds; CBCL; Achenbach & Rescorla, 2000). Parents will complete this widely used 100-item questionnaire to report their children's internalizing (36 items, e.g., "is nervous, withdrawn") and externalizing (24 items, e.g., "is restless, disobedient") behavior problems. Responses are given on a 3-point scale: (0) not true, (1). somewhat/ sometimes true, (2) very/often true). Items are summed to create subscales for internalizing and externalizing problems.
Child Behavior Checklist (CBCL) #3 | 6-month follow up
  Child behavior problems will are assessed with the Child Behavior Checklist (version for 1.5- to 5-year-olds; CBCL; Achenbach & Rescorla, 2000). Parents will complete this widely used 100-item questionnaire to report their children's internalizing (36 items, e.g., "is nervous, withdrawn") and externalizing (24 items, e.g., "is restless, disobedient") behavior problems. Responses are given on a 3-point scale: (0) not true, (1). somewhat/ sometimes true, (2) very/often true). Items are summed to create subscales for internalizing and externalizing problems.
Infant-Toddler Social and Emotional Assessment (ITSEA) #1 | Baseline
  Child behavior problems (from parent report) will be assessed with the ITSEA (Carter & Briggs-Gowan, 2000; Carter et al., 2003) for children below the age of 1.5 years. The ITSEA assesses internalizing and externalizing symptoms. Parents will rate items on a scale of 0 (not true) to 2 (very true).
Infant-Toddler Social and Emotional Assessment (ITSEA) #2 | Immediately post-intervention
  Child behavior problems (from parent report) will be assessed with the ITSEA (Carter & Briggs-Gowan, 2000; Carter et al., 2003) for children below the age of 1.5 years. The ITSEA assesses internalizing and externalizing symptoms. Parents will rate items on a scale of 0 (not true) to 2 (very true).
Infant-Toddler Social and Emotional Assessment (ITSEA) #3 | 6-month follow up
  Child behavior problems (from parent report) will be assessed with the ITSEA (Carter & Briggs-Gowan, 2000; Carter et al., 2003) for children below the age of 1.5 years. The ITSEA assesses internalizing and externalizing symptoms. Parents will rate items on a scale of 0 (not true) to 2 (very true).
Parental Emotional Responses to Child Distress #1 | Baseline
  Parental emotional response to child distress will be assessed with the Crying Infant Video Task (Leerkes et al., 2004, 2011), in which parents watch four one-minute videos of (gender-neutral, racially diverse) infants in distress (i.e., crying loudly and continuously while sitting in a highchair). Following each clip, parents complete a questionnaire (4-point scale; 17 items) about their emotions while watching the clips, and elaborate about these emotions. Mean intensity scores are used to create a child-oriented empathic emotional response score (e.g., child-oriented sad, sympathy) and a parent-oriented negative emotions score (e.g., parent-oriented irritated, angry; see Leerkes, 2010).
Parental Emotional Responses to Child Distress #2 | Immediately post-intervention
  Parental emotional response to child distress will be assessed with the Crying Infant Video Task (Leerkes et al., 2004, 2011), in which parents watch four one-minute videos of (gender-neutral, racially diverse) infants in distress (i.e., crying loudly and continuously while sitting in a highchair). Following each clip, parents complete a questionnaire (4-point scale; 17 items) about their emotions while watching the clips, and elaborate about these emotions. Mean intensity scores are used to create a child-oriented empathic emotional response score (e.g., child-oriented sad, sympathy) and a parent-oriented negative emotions score (e.g., parent-oriented irritated, angry; see Leerkes, 2010).
Parental Emotional Responses to Child Distress #3 | 6-month follow up
  Parental emotional response to child distress will be assessed with the Crying Infant Video Task (Leerkes et al., 2004, 2011), in which parents watch four one-minute videos of (gender-neutral, racially diverse) infants in distress (i.e., crying loudly and continuously while sitting in a highchair). Following each clip, parents complete a questionnaire (4-point scale; 17 items) about their emotions while watching the clips, and elaborate about these emotions. Mean intensity scores are used to create a child-oriented empathic emotional response score (e.g., child-oriented sad, sympathy) and a parent-oriented negative emotions score (e.g., parent-oriented irritated, angry; see Leerkes, 2010).
Electrodermal Activity (EDA) arousal #1 | Baseline
  Parental EDA arousal in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA). For EDA investigators will attach two silver chloride electrodes to the palmar surface of the second phalanges of the index and middle fingers of each participant's non-dominant hand. EDA sample rate will be 1000 samples per second. Phasic skin conductance will be calculated using a smoothing filter with a window width of 0.25 seconds. Skin conductance responses (SCRs) will be calculated using a threshold of 0.05 µS. The EDA variable will be the sum the SCRs across the four videos.
Electrodermal Activity (EDA) arousal #2 | Immediately post-intervention
  Parental EDA arousal in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA). For EDA investigators will attach two silver chloride electrodes to the palmar surface of the second phalanges of the index and middle fingers of each participant's non-dominant hand. EDA sample rate will be 1000 samples per second. Phasic skin conductance will be calculated using a smoothing filter with a window width of 0.25 seconds. Skin conductance responses (SCRs) will be calculated using a threshold of 0.05 µS. The EDA variable will be the sum the SCRs across the four videos.
Electrodermal Activity (EDA) arousal #3 | 6-month follow up
  Parental EDA arousal in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA). For EDA investigators will attach two silver chloride electrodes to the palmar surface of the second phalanges of the index and middle fingers of each participant's non-dominant hand. EDA sample rate will be 1000 samples per second. Phasic skin conductance will be calculated using a smoothing filter with a window width of 0.25 seconds. Skin conductance responses (SCRs) will be calculated using a threshold of 0.05 µS. The EDA variable will be the sum the SCRs across the four videos.
Respiratory Sinus Arrhythmia (RSA) #1 | Baseline
  Parental RSA change in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA) and respiratory sinus arrhythmia (RSA). For RSA, investigators will attach three electrodes in a modified Lead II placement on the distal end of the right clavicle, lower left rib cage chest, and right rib cage of each parent's chest. The ECG signal will be sampled continuously with low-pass filtering at 1000 Hertz and passed through an Analog-to-Digital converter. RSA values will be derived from the interbeat interval series and resampled at 25 msec to create a stationary wave form. The integral of the power in the RSA band (0.12 to 0.40 for parents) will be extracted to obtain the RSA statistics in 30-second epochs, and will be used to calculate RSA change in response to infant distress.
Respiratory Sinus Arrhythmia (RSA) #2 | Immediately post-intervention
  Parental RSA change in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA) and respiratory sinus arrhythmia (RSA). For RSA, investigators will attach three electrodes in a modified Lead II placement on the distal end of the right clavicle, lower left rib cage chest, and right rib cage of each parent's chest. The ECG signal will be sampled continuously with low-pass filtering at 1000 Hertz and passed through an Analog-to-Digital converter. RSA values will be derived from the interbeat interval series and resampled at 25 msec to create a stationary wave form. The integral of the power in the RSA band (0.12 to 0.40 for parents) will be extracted to obtain the RSA statistics in 30-second epochs, and will be used to calculate RSA change in response to infant distress.
Respiratory Sinus Arrhythmia (RSA) #3 | 6-month follow up
  Parental RSA change in response to child distress will be assessed during the Crying Infant Video Task (above). Investigators will use a MindWare BioNex 8-Slot Chassis Assembly and BioLab Acquisition Software to tap parental electrodermal activity (EDA) and respiratory sinus arrhythmia (RSA). For RSA, investigators will attach three electrodes in a modified Lead II placement on the distal end of the right clavicle, lower left rib cage chest, and right rib cage of each parent's chest. The ECG signal will be sampled continuously with low-pass filtering at 1000 Hertz and passed through an Analog-to-Digital converter. RSA values will be derived from the interbeat interval series and resampled at 25 msec to create a stationary wave form. The integral of the power in the RSA band (0.12 to 0.40 for parents) will be extracted to obtain the RSA statistics in 30-second epochs, and will be used to calculate RSA change in response to infant distress.
Coping with Toddlers' Negative Emotions Scale (CTNES) #1 | Baseline
  Parental behavioral sensitivity in response to child distress will be assessed using the Coping With Toddlers' Negative Emotions Scale (CTNES; Spinrad et al., 2007), parents will report their likely behavior on a scale of 1 (very likely) to 7 (very unlikely) in response to 12 hypothetical situations with their distressed child (e.g., "If my child becomes upset and cries because he is left alone…, I would:"). For each item, parents report their likelihood of responding in six different ways, for instance punitive responses (i.e., punishing the child); minimizing responses (i.e., telling child to stop overreacting); emotion-focused reactions (i.e., comforting); and problem-focused reactions (i.e., helping child come up with solution). Following Gudmundson and Leerkes (2012), investigators will form supportive and unsupportive parental response composites.
Coping with Toddlers' Negative Emotions Scale (CTNES) #2 | Immediately post-intervention
  Parental behavioral sensitivity in response to child distress will be assessed using the Coping With Toddlers' Negative Emotions Scale (CTNES; Spinrad et al., 2007), parents will report their likely behavior on a scale of 1 (very likely) to 7 (very unlikely) in response to 12 hypothetical situations with their distressed child (e.g., "If my child becomes upset and cries because he is left alone…, I would:"). For each item, parents report their likelihood of responding in six different ways, for instance punitive responses (i.e., punishing the child); minimizing responses (i.e., telling child to stop overreacting); emotion-focused reactions (i.e., comforting); and problem-focused reactions (i.e., helping child come up with solution). Following Gudmundson and Leerkes (2012), investigators will form supportive and unsupportive parental response composites.
Coping with Toddlers' Negative Emotions Scale (CTNES) #3 | 6 month follow up
  Parental behavioral sensitivity in response to child distress will be assessed using the Coping With Toddlers' Negative Emotions Scale (CTNES; Spinrad et al., 2007), parents will report their likely behavior on a scale of 1 (very likely) to 7 (very unlikely) in response to 12 hypothetical situations with their distressed child (e.g., "If my child becomes upset and cries because he is left alone…, I would:"). For each item, parents report their likelihood of responding in six different ways, for instance punitive responses (i.e., punishing the child); minimizing responses (i.e., telling child to stop overreacting); emotion-focused reactions (i.e., comforting); and problem-focused reactions (i.e., helping child come up with solution). Following Gudmundson and Leerkes (2012), investigators will form supportive and unsupportive parental response composites.
Stranger Approach Lab-TAB Task to Assess Parental Behavioral Sensitivity #1 | Baseline
  Raters will observe parental behavioral sensitivity during the 'Stranger Approach' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit fearfulness in children by having an adult stranger approach the child. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.
Jar Lab-TAB Task to Assess Parental Behavioral Sensitivity #1 | Baseline
  Raters will observe parental behavioral sensitivity during the 'Jar' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit frustration and anger in children by placing an attractive snack (e.g. rainbow goldfish), in a plastic jar. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.
Stranger Approach Lab-TAB Task to Assess Parental Behavioral Sensitivity #2 | Immediately post-intervention
  Raters will observe parental behavioral sensitivity during the 'Stranger Approach' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit fearfulness in children by having an adult stranger approach the child. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.
Jar Lab-TAB Task to Assess Parental Behavioral Sensitivity #2 | Immediately post-intervention
  Raters will observe parental behavioral sensitivity during the 'Jar' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit frustration and anger in children by placing an attractive snack (e.g. rainbow goldfish), in a plastic jar. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.
Stranger Approach Lab-TAB Task to Assess Parental Behavioral Sensitivity #3 | 6-month follow up
  Raters will observe parental behavioral sensitivity during the 'Stranger Approach' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit fearfulness in children by having an adult stranger approach the child. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.
Jar Lab-TAB Task to Assess Parental Behavioral Sensitivity #3 | 6-month follow up
  Raters will observe parental behavioral sensitivity during the 'Jar' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit frustration and anger in children by placing an attractive snack (e.g. rainbow goldfish), in a plastic jar. This task lasts less than 2 minutes. The first 2 minutes are coded for child temperament, with 5 minutes then coded for parental sensitivity. Given the investigators' particular focus to sensitivity to distress, investigators will retain their analytic focus on sensitivity during distress, yet collection of both will allow for additional exploratory analyses in the future. Parental sensitivity (4-point scale) will be coded following the National Institute of Child Health and and Human Development (NICHD; 1999) guidelines.

SECONDARY OUTCOMES:
Financial Stress Questionnaire #1 | Baseline
  The Financial Stress Questionnaire is a 9-item instrument, developed by the Fast Track project (CPPRG, 1994), which explores sources of household spending and adequacy of funds for paying bills. The questionnaire is administered to parents. The parent is asked to evaluate the affordability of 7 spending sources in the household (home, clothing, furniture, car, food, medical care and leisure) on a 1 to 5 scale (strongly agree, agree, neutral, disagree, strongly disagree); how much difficulty he/she had to pay the bills on a 1 to 5 scale (a great of difficulty to no difficulty at all) and how much money was left at the end of the month on a 1 to 4 scale (not enough, just enough, some money left, more than enough money left over).
Financial Stress Questionnaire #2 | Immediately post-intervention
  The Financial Stress Questionnaire is a 9-item instrument, developed by the Fast Track project (CPPRG, 1994), which explores sources of household spending and adequacy of funds for paying bills. The questionnaire is administered to parents. The parent is asked to evaluate the affordability of 7 spending sources in the household (home, clothing, furniture, car, food, medical care and leisure) on a 1 to 5 scale (strongly agree, agree, neutral, disagree, strongly disagree); how much difficulty he/she had to pay the bills on a 1 to 5 scale (a great of difficulty to no difficulty at all) and how much money was left at the end of the month on a 1 to 4 scale (not enough, just enough, some money left, more than enough money left over).
Financial Stress Questionnaire #3 | 6-month follow-up
  The Financial Stress Questionnaire is a 9-item instrument, developed by the Fast Track project (CPPRG, 1994), which explores sources of household spending and adequacy of funds for paying bills. The questionnaire is administered to parents. The parent is asked to evaluate the affordability of 7 spending sources in the household (home, clothing, furniture, car, food, medical care and leisure) on a 1 to 5 scale (strongly agree, agree, neutral, disagree, strongly disagree); how much difficulty he/she had to pay the bills on a 1 to 5 scale (a great of difficulty to no difficulty at all) and how much money was left at the end of the month on a 1 to 4 scale (not enough, just enough, some money left, more than enough money left over).
O'Leary-Porter Overt Hostility Scale #1 | Baseline
  Marital Stress will be assessed using the 10-item O'Leary-Porter Overt Hostility Scale, which measures how often parents openly argue, display physical and verbal hostility, and criticize each other in the presence of the children (Johnson & O'Leary, 1987; Porter & O'Leary, 1980). The scale uses a 6-point scale from 1 = never to 6 = very often. Investigators made slight modifications to this scale to reduce the focus on only marital relationships. Participants under 20 years of age will receive a 9-item version of this scale to avoid asking younger participants about experiences of witnessing physical violence.
O'Leary-Porter Overt Hostility Scale #2 | Immediately post-intervention
  Marital Stress will be assessed using the 10-item O'Leary-Porter Overt Hostility Scale, which measures how often parents openly argue, display physical and verbal hostility, and criticize each other in the presence of the children (Johnson & O'Leary, 1987; Porter & O'Leary, 1980). The scale uses a 6-point scale from 1 = never to 6 = very often. Investigators made slight modifications to this scale to reduce the focus on only marital relationships. Participants under 20 years of age will receive a 9-item version of this scale to avoid asking younger participants about experiences of witnessing physical violence.
O'Leary-Porter Overt Hostility Scale #3 | 6-month follow-up
  Marital Stress will be assessed using the 10-item O'Leary-Porter Overt Hostility Scale, which measures how often parents openly argue, display physical and verbal hostility, and criticize each other in the presence of the children (Johnson & O'Leary, 1987; Porter & O'Leary, 1980). The scale uses a 6-point scale from 1 = never to 6 = very often. Investigators made slight modifications to this scale to reduce the focus on only marital relationships. Participants under 20 years of age will receive a 9-item version of this scale to avoid asking younger participants about experiences of witnessing physical violence.
Adverse Childhood Experiences Questionnaire (ACE-Q) | Baseline
  The Adverse Childhood Experience Questionnaire (ACE-Q; Felitti et al., 1998) is a brief rating scale that measures the number of adverse childhood experiences that occurred in the first 18 years of life. The ACE-Q has 9 yes/no items that count the number of adverse childhood experiences participants experienced in the first 18 years of their life. A sample item is "Did a parent or other adult in the household often swear at you, insult you, put you down, or humiliate you? OR act in a way that made you afraid that you might be physically hurt?" Participants indicate yes or no for each question, and if the answer is yes, then a score of 1 is entered for that item. The number of ACEs is the total number of questions for which the answer was yes. To avoid asking younger participants about experiences of physical or sexual abuse, this questionnaire will only be given to participants over 20 years of age.
Role Overload #1 | Baseline
  Following the recommendations of Thiagarajan et al. (2006), Reilly's (1982) 13-item Role Overload Scale will be adapted into a 6-item unidimensional scale assessing parents' feelings of being overwhelmed with parenting duties, juggling multiple obligations, and lacking time to rest or pursue desired activities (e.g., "I cannot ever seem to catch up"). Parents' scores indicating how often they agree with the corresponding statements, using a 7-point scale which ranges from 1 = Never to 7 = Always, will be averaged.
Role Overload #2 | Immediately post-intervention
  Following the recommendations of Thiagarajan et al. (2006), Reilly's (1982) 13-item Role Overload Scale will be adapted into a 6-item unidimensional scale assessing parents' feelings of being overwhelmed with parenting duties, juggling multiple obligations, and lacking time to rest or pursue desired activities (e.g., "I cannot ever seem to catch up"). Parents' scores indicating how often they agree with the corresponding statements, using a 7-point scale which ranges from 1 = Never to 7 = Always, will be averaged.
Role Overload #3 | 6-month follow-up
  Following the recommendations of Thiagarajan et al. (2006), Reilly's (1982) 13-item Role Overload Scale will be adapted into a 6-item unidimensional scale assessing parents' feelings of being overwhelmed with parenting duties, juggling multiple obligations, and lacking time to rest or pursue desired activities (e.g., "I cannot ever seem to catch up"). Parents' scores indicating how often they agree with the corresponding statements, using a 7-point scale which ranges from 1 = Never to 7 = Always, will be averaged.
My Exposure to Violence | Baseline
  Witnessing community violence and violent victimization will be assessed using two subscales (victimization and witnessing) of the My Exposure to Violence (MyETV; Selner-O'Hagan et al., 1998). This is a 25-item instrument that was designed to measure participants' exposure to violence in the past year. The MyETV asks participants about witnessed as well as personally experienced violence, yielding three subscales (of which investigators will use two). The three subscales are witnessing violence, violent victimization, and total exposure. Frequency of exposure is measured on a 4-point scale (once, 2 or 3 times, 4 to 10 times, more than 10 times). To avoid asking questions about childhood physical or sexual abuse, this questionnaire will only be given to participants over 20 years of age.
Experiences in Close Relationships Scale (ECR) #1 | Baseline
  Adult attachment style will be assessed with the 36-item self-report Experiences in Close Relationships Scale (ECR; Brennan, Clark, & Shaver, 1998; see Mikulincer & Shaver, 2016). The ECR assesses two dimensions of adult attachment style: attachment related avoidance (discomfort with closeness and intimacy) and attachment related anxiety (intense fear of rejection and abandonment) each on a scale of 1 (low) to 7 (high).
Experiences in Close Relationships Scale (ECR) #2 | Immediately post-intervention
  Adult attachment style will be assessed with the 36-item self-report Experiences in Close Relationships Scale (ECR; Brennan, Clark, & Shaver, 1998; see Mikulincer & Shaver, 2016). The ECR assesses two dimensions of adult attachment style: attachment related avoidance (discomfort with closeness and intimacy) and attachment related anxiety (intense fear of rejection and abandonment) each on a scale of 1 (low) to 7 (high).
Experiences in Close Relationships Scale (ECR) #3 | 6-month follow-up
  Adult attachment style will be assessed with the 36-item self-report Experiences in Close Relationships Scale (ECR; Brennan, Clark, & Shaver, 1998; see Mikulincer & Shaver, 2016). The ECR assesses two dimensions of adult attachment style: attachment related avoidance (discomfort with closeness and intimacy) and attachment related anxiety (intense fear of rejection and abandonment) each on a scale of 1 (low) to 7 (high).
Center for Epidemiologic Studies Depression Scale (CES-D) #1 | Baseline
  Parental depressive symptoms will be assessed with the CES-D (Radloff, 1977). This 20-item self-report measure (Radloff, 1977) taps the frequency with which respondents experienced depressive symptoms over the past week. Responses are given on a 4-point scale, with 0 indicating that the symptom was rarely or never felt, and 3 indicating that it was experienced most or all of the time.
Center for Epidemiologic Studies Depression Scale (CES-D) #2 | Immediately post-intervention
  Parental depressive symptoms will be assessed with the CES-D (Radloff, 1977). This 20-item self-report measure (Radloff, 1977) taps the frequency with which respondents experienced depressive symptoms over the past week. Responses are given on a 4-point scale, with 0 indicating that the symptom was rarely or never felt, and 3 indicating that it was experienced most or all of the time.
Center for Epidemiologic Studies Depression Scale (CES-D) #3 | 6-month follow-up
  Parental depressive symptoms will be assessed with the CES-D (Radloff, 1977). This 20-item self-report measure (Radloff, 1977) taps the frequency with which respondents experienced depressive symptoms over the past week. Responses are given on a 4-point scale, with 0 indicating that the symptom was rarely or never felt, and 3 indicating that it was experienced most or all of the time.
Child Behavior Questionnaire | Baseline
  Parents will complete the age appropriate version of the Child Behavior Questionnaires designed by Rothbart & colleagues (e.g., Putnam & Rothbart, 2006). This questionnaire assesses child temperamental reactivity and child fearful temperament.
Stranger Approach Lab-TAB Task to assess child temperament | Baseline
  Raters will observe child temperament during the 'Stranger Approach' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit fearfulness by having an adult stranger approach and stare at the child in a standardized fashion. The elements of novelty and intrusiveness should elicit various degrees of fearful distress and avoidance. This task lasts approximately 1-2 minutes.
Behind Barrier Lab-TAB Task to assess child temperament | Baseline
  Raters will observe child temperament during the 'Behind Barrier' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit frustration and anger by placing a toy, with which the child has been playing, behind a barrier. Anger is coded as verbal and physical action against the barrier or persons present. This task lasts approximately 3 minutes.
Jar Lab-TAB Task to assess child temperament | Baseline
  Raters will observe child temperament during the 'Jar' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit frustration and anger by placing an attractive snack (e.g. rainbow goldfish), in a plastic jar. This action is representative of the type of frustration a child typically encounters when exploration or play is blocked. Anger is coded as verbal and physical action against the jar or persons present. This task lasts approximately 1-2 minutes.
Spider Lab-TAB Task to assess child temperament | Baseline
  Raters will observe child temperament during the 'Spider' Lab-TAB task (Goldsmith & Rothbart, 1999), a task designed to elicit fearfulness by having a toy spider unexpectedly approach the child. The elements of novelty, uncertainty and intrusiveness, as well as a possible fear of animals, should elicit varying degrees of fear. This task lasts approximately 2-3 minutes.
Infant Behavior Record (IBR) assessing child temperament #1 | Baseline
  Two trained observers will use the Infant Behavior Record (IBR; Bayley, 1969; Stifter & Corey, 2001; Stifter et al., 2008) to assess 11 dimensions of child temperament based on their observations of the entire lab session.
Infant Behavior Record (IBR) assessing child temperament #2 | Immediately post-intervention
  Two trained observers will use the Infant Behavior Record (IBR; Bayley, 1969; Stifter & Corey, 2001; Stifter et al., 2008) to assess 11 dimensions of child temperament based on their observations of the entire lab session.
Infant Behavior Record (IBR) assessing child temperament #3 | 6-month follow-up
  Two trained observers will use the Infant Behavior Record (IBR; Bayley, 1969; Stifter & Corey, 2001; Stifter et al., 2008) to assess 11 dimensions of child temperament based on their observations of the entire lab session.
Experience of Discrimination Scale (EOD) | Baseline
  Participants' lifetime experience with discrimination will be assessed using the 9-item self-report Experience of Discrimination Scale (EOD; Krieger, 1990; Krieger & Sidney, 1996; Krieger et al., 2005). Following Krieger et al. (2005), investigators included an additional 4 questions about participants' level of worry about experiencing unfair treatment due to their race or ethnicity.

OTHER OUTCOMES:
Parent-Reported Demographic Variables #1 | Baseline
  Demographic variables are parent age, education, occupation, language(s) spoken, number of children, people living in the household, relationship status, single/living with partner, family income, racial/ethnic identity, enrollment status in Early Head Starts, experience of homelessness, whether they receive benefits from Temporary Assistance for Needy Families or Supplemental Security Income, as well as the target child's age, sex, race/ethnicity, childcare, whether the child was born prematurely, and autism diagnosis.
Parent-Reported Demographic Variables #2 | Immediately post-intervention
  Immediately post-intervention, caregivers will answer a selected set of demographic variables including their occupation, number of children, people living in the household, relationship status, and autism diagnosis.
Parent-Reported Demographic Variables #3 | 6-month follow-up
  At the 6-month follow-up, caregivers will answer a selected set of demographic variables including their occupation, number of children, people living in the household, relationship status, and autism diagnosis.
Observer Ratings of Intervener Treatment Adherence and Competence for COS-P | From COS-P intervention onset to completion, 8 weeks
  All sessions will be videotaped. Investigators will code a randomly selected 20 percent of Circle of Security Parenting (COS-P) sessions (stratified by intervener) to be coded (with a 30 percent reliability overlap) by independent blind coders for treatment adherence and intervener competence using a COS-P-specific adaptation of the Yale Adherence and Competence Scale (YACS; Carroll et al., 2000). Each session will be coded for COS-P-specific items on two dimensions: Adherence (1 = not at all, 7 = extensively) and Skill Level (competence with which the intervener delivered specific aspects of the intervention, 1 = very poor, 7 = excellent). Items reflect specific manualized content (e.g., COS-P model for understanding child needs) and process (e.g., supporting parent observation skills, building a strong alliance). Scores of competence that are = or > 3 reflect sufficient to excellent competence, whereas scores < 3 reflect lack of competence.
Observer Ratings of Intervener Treatment Adherence and Competence for Little Talks | From Little Talks intervention onset to completion, 8 weeks
  Investigators will code a randomly selected 20 percent of sessions (stratified by intervener) to be coded (with a 30 percent reliability overlap) by independent masked coders for intervener adherence/competence using the Little Talks Fidelity Form (Manz et al., 2017). The Little Talks Fidelity form reflects the specific manualized content of Little Talks in four categories: Little Talks Curriculum fidelity (6 items), Collaborative Goal Setting fidelity (6 items), Home Visitor Decision Making fidelity (2 items), and Parent Collaboration fidelity (6 items). Each item is scored as either 1 = delivered with sufficient competency or 0 = not delivered with sufficient competency. For the purpose of comparing Little Talks intervener competence with COS-P intervener competence, Little Talks Fidelity scores can be used to create a score representing percentage of intervention delivered with sufficient competence (total number of items = 1 / total number of items).
COS-P Intervener Adherence Checklist | From COS-P intervention onset to completion, 8 weeks
  For adherence, interveners will complete a checklist at the end of each session indicating whether or not they accomplished the session goals as outlined in the manual, as well as a standardized COS-P session journal that asks interveners to reflect in writing on two specific instances from the session in which they dealt with particular topics. The fidelity team will review completed checklists and journals weekly to monitor intervention component completion and so prevent implementation drift. Specifically, the fidelity team will monitor whether all components were completed, and alert the intervener to cover any absent material the following week; the following week's session will then be reviewed to ensure the material was covered. The checklist includes both content and process items.
Little Talks Intervener Fidelity form (Intervener Rated) | From Little Talks intervention onset to completion, 8 weeks
  For adherence, interveners will complete the Little Talks Intervener Fidelity form (Manz et al., 2017) at the end of each session. The Little Talks Fidelity form reflects the specific manualized content of Little Talks in four categories: Little Talks Curriculum fidelity (6 items), Collaborative Goal Setting fidelity (6 items), Home Visitor Decision Making fidelity (2 items), and Parent Collaboration fidelity (6 items). Each item is scored as either 1 = delivered with sufficient competency or 0 = not delivered with sufficient competency.
Participant Ratings of Intervener Competence | Immediately post-intervention (for both COS-P & Little Talks)
  Participants will rate their interveners' competence as part of the post-intervention lab assessment using the 12-item Counselor Rating Form-Short (CRF-S; Corrigan & Schmidt, 1983; Wilson & Yager, 1990). Participants in each intervention group (COS-P & Little Talks) will complete these ratings. Participants will rate how much the intervener displays characteristics (e.g., "friendly," "reliable," "prepared") on a scale of 1 (not very) to 7 (very). The CRF-S is a general measure of client perceptions of intervener competence.
Participant Ratings of Intervention Service | Immediately post-intervention (for both COS-P & Little Talks)
  Participant evaluations of the intervention service (Carroll et al., 2007) will be gathered using the widely used (participant-reported) Client Satisfaction Questionnaire (CSQ-8; Nguyen et al., 1983). Participants in each intervention group (COS-P & Little Talks) will complete these ratings. Participants will answer questions about their satisfaction with the service on a 4-point scale (1 reflecting poorer satisfaction, 4 reflecting higher satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Jude Cassidy, Ph.D., Principal Investigator — University of Maryland, College Park; Susan Woodhouse, Ph.D., Principal Investigator — Lehigh University
Locations (2):
- United States (2):
  - University of Maryland, College Park, College Park, Maryland
  - Lehigh University, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Achenbach, T. M., & Rescorla, L. A. (2000). Manual for the ASEBA Preschool Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Ainsworth, M., Blehar, M., Waters, E., & Wall, S. (1978). Patterns of attachment. Erlbaum.
- [Background] Bayley, N. 1969. Bayley scales of infant development. New York: Psychological Corp.
- [Background] Bernard K, Dozier M. Examining infants' cortisol responses to laboratory tasks among children varying in attachment disorganization: stress reactivity or return to baseline? Dev Psychol. 2010 Nov;46(6):1771-8. doi: 10.1037/a0020660. PMID 20873923
- [Background] Bowlby, J. (1988). A secure base. Basic Books.
- [Background] Brennan, K. A., Clark, C. L., & Shaver, P. R. (1998). Self-report measurement of adult attachment: An integrative overview. In J. A. Simpson, W. S. Rholes, J. A. Simpson, W. S. Rholes (Eds.), Attachment theory and close relationships (pp. 46-76). Guilford.
- [Background] Carroll KM, Nich C, Sifry RL, Nuro KF, Frankforter TL, Ball SA, Fenton L, Rounsaville BJ. A general system for evaluating therapist adherence and competence in psychotherapy research in the addictions. Drug Alcohol Depend. 2000 Jan 1;57(3):225-38. doi: 10.1016/s0376-8716(99)00049-6. PMID 10661673
- [Background] Carter, A. S., & Briggs-Gowan, M. J. (2000). The Infant-Toddler Social and Emotional Assessment (ITSEA). Unpublished Manual. University of Massachusetts Boston Department of Psychology, Boston, MA. Yale University, New Haven, CT. Available by request at alice.carter@umb.edu.
- [Background] Carter AS, Briggs-Gowan MJ, Jones SM, Little TD. The Infant-Toddler Social and Emotional Assessment (ITSEA): factor structure, reliability, and validity. J Abnorm Child Psychol. 2003 Oct;31(5):495-514. doi: 10.1023/a:1025449031360. PMID 14561058
- [Background] Cassidy, J., & Marvin, R. S., with MacArthur Attachment Working Group (1992). Attachment organization in preschool children: Procedures and coding manual (4th ed.). Unpublished manuscript, Department of Psychology, University of Virginia, Charlottesville, Virginia.
- [Background] Conduct Problems Prevention Research Group (CPPRG). (1994). Financial Stress Questionnaire. Available from the Fast Track Project Web site: http://www.fasttrackproject.org
- [Background] Corrigan, J., & Schmidt, L. (1983). Development and validation of revisions in the Counselor Rating Form. Journal of Counseling Psychology, 30, 64-75. doi: 10.1037/0022-0167.30.1.64
- [Background] Felitti, V. J., Anda, R. F., Nordenberg, D., & Williamson, D. F. (1998). Adverse childhood experiences and health outcomes in adults: The Ace study. Journal of Family and Consumer Sciences, 90, 31.
- [Background] Goldsmith, H. H., & Rothbart, M. K. (1999). The Laboratory Temperament Assessment Battery. Locomotor Version 3.1, Description of Procedures. University of Wisconsin, Madison, WI.
- [Background] Gudmundson JA, Leerkes EM. Links between mothers' coping styles, toddler reactivity, and sensitivity to toddler's negative emotions. Infant Behav Dev. 2012 Feb;35(1):158-66. doi: 10.1016/j.infbeh.2011.07.004. Epub 2011 Sep 7. PMID 21903276
- [Background] Gunnar, M. R., & Herrera, A. M. (2013). The development of stress reactivity: A neurobiological perspective. In P. D. Zelazo (Ed.), The Oxford handbook of developmental psychology, Vol. 2. Self and other (pp. 45-80). Oxford University Press.
- [Background] Johnson PL, O'Leary KD. Parental behavior patterns and conduct disorders in girls. J Abnorm Child Psychol. 1987 Dec;15(4):573-81. doi: 10.1007/BF00917242. PMID 3437092
- [Background] Krieger N. Racial and gender discrimination: risk factors for high blood pressure? Soc Sci Med. 1990;30(12):1273-81. doi: 10.1016/0277-9536(90)90307-e. PMID 2367873
- [Background] Krieger N, Sidney S. Racial discrimination and blood pressure: the CARDIA Study of young black and white adults. Am J Public Health. 1996 Oct;86(10):1370-8. doi: 10.2105/ajph.86.10.1370. PMID 8876504
- [Background] Krieger N, Smith K, Naishadham D, Hartman C, Barbeau EM. Experiences of discrimination: validity and reliability of a self-report measure for population health research on racism and health. Soc Sci Med. 2005 Oct;61(7):1576-96. doi: 10.1016/j.socscimed.2005.03.006. Epub 2005 Apr 21. PMID 16005789
- [Background] Leerkes EM. Predictors of Maternal Sensitivity to Infant Distress. Parent Sci Pract. 2010 Jul 1;10(3):219-239. doi: 10.1080/15295190903290840. PMID 20824194
- [Background] Leerkes, E. M., Crockenberg, S. C., & Burrous, E. (2004). Identifying components of maternal sensitivity to infant distress: The role of maternal emotional competencies. Parenting: Science and Practice, 4, 1-23. doi:10.1207/s15327922par04011
- [Background] Leerkes EM, Parade SH, Gudmundson JA. Mothers' emotional reactions to crying pose risk for subsequent attachment insecurity. J Fam Psychol. 2011 Oct;25(5):635-43. doi: 10.1037/a0023654. PMID 21517171
- [Background] Luijk MP, Saridjan N, Tharner A, van Ijzendoorn MH, Bakermans-Kranenburg MJ, Jaddoe VW, Hofman A, Verhulst FC, Tiemeier H. Attachment, depression, and cortisol: Deviant patterns in insecure-resistant and disorganized infants. Dev Psychobiol. 2010 Jul;52(5):441-52. doi: 10.1002/dev.20446. PMID 20583141
- [Background] Manz, P. H., Eisenberg, R., Gernhart, A., Faison, J., Laracy, S., Ridgard, T. & Pinho, T. (2016). Engaging Early Head Start parents in a collaborative inquiry: The co-construction of Little Talks, Early Child Development and Care. doi: 10.1080/03004430.2016.1169177
- [Background] Manz, P. H., Power, T. J., Roggman, L. A., Eisenberg, R. A., Gernhart, A., Faison, J., Ridgard, T., Wallace, L. E., & Whitenack, J. M. (2017). Integrating the Little Talks intervention into Early Head Start: An experimental examination of implementation supports involving fidelity monitoring and performance feedback. Children and Youth Services Review, 79, 87-96. doi 10.1016/j.childyouth.2017.05.034
- [Background] Mikulincer, M., & Shaver, P. R. (2016). Attachment in adulthood: Structure, dynamics, and change (2nd ed.). Guilford.
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Child care and mother-child interaction in the first 3 years of life. NICHD Early Child Care Research Network. Dev Psychol. 1999 Nov;35(6):1399-413. PMID 10563730
- [Background] Porter B, O'Leary KD. Marital discord and childhood behavior problems. J Abnorm Child Psychol. 1980 Sep;8(3):287-95. doi: 10.1007/BF00916376. PMID 7410730
- [Background] Putnam SP, Rothbart MK. Development of short and very short forms of the Children's Behavior Questionnaire. J Pers Assess. 2006 Aug;87(1):102-12. doi: 10.1207/s15327752jpa8701_09. PMID 16856791
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1, 385-401. doi: 10.1177/014662167700100306
- [Background] Reilly, M. D. (1982). Working wives and convenience consumption. Journal of Consumer Research, 8(4), 407-418. https://doi.org/10.1086/208881
- [Background] Selner-O'Hagan MB, Kindlon DJ, Buka SL, Raudenbush SW, Earls FJ. Assessing exposure to violence in urban youth. J Child Psychol Psychiatry. 1998 Feb;39(2):215-24. PMID 9669234
- [Background] Solomon, J., & George, C. (2016). The measurement of attachment security and related constructs in infancy and early childhood. In J. Cassidy & P. R. Shaver (Eds.), Handbook of attachment: Theory, research, and clinical applications (3rd ed., pp. 366-398). Guilford.
- [Background] Spinrad TL, Eisenberg N, Gaertner B, Popp T, Smith CL, Kupfer A, Greving K, Liew J, Hofer C. Relations of maternal socialization and toddlers' effortful control to children's adjustment and social competence. Dev Psychol. 2007 Sep;43(5):1170-86. doi: 10.1037/0012-1649.43.5.1170. PMID 17723043
- [Background] Stifter, C. A., & Corey, J. M. (2001). Vagal regulation and observed social behavior in infancy. Social Development, 10(2), 189-201. https://doi.org/10.1111/1467-9507.00158
- [Background] Stifter CA, Willoughby MT, Towe-Goodman N; The Family Life Project Key Investigators. Agree or Agree to Disagree? Assessing the Convergence between Parents and Observers on Infant Temperament. Infant Child Dev. 2008 Aug 1;17(4):407-426. doi: 10.1002/icd.584. PMID 19936035
- [Background] Thiagarajan, P., Chakrabarty, S., & Taylor, R. D. (2006). A confirmatory factor analysis of Reilly's Role Overload Scale. Educational and Psychological Measurement, 66(4), 657-666. https://doi.org/10.1177/0013164405282452
- [Background] Thompson LA, Morgan G, Jurado KA, Gunnar MR. III. JUSTIFICATION FOR CORTISOL RESPONSE CATEGORIES. Monogr Soc Res Child Dev. 2015 Dec;80(4):40-7. doi: 10.1111/mono.12210. No abstract available. PMID 26496583
- [Background] Wilson, F., & Yager, G. (1990). Concurrent and construct validity of three counselor social influence instruments. Measurement and Evaluation in Counseling and Development, 23, 52-66.